CLINICAL TRIAL: NCT01193465
Title: Comparison of Heat and Humidity Conservation Among Different Anesthesia Workstation and Different Flow Rate.
Brief Title: Temperature and Humidity Among Different Anesthesia Work-station
Acronym: humidity
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Seung Zhoo Yoon, Department of anesthesiology and pain medicine Korea University Anam Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: humidity
Record Dates: First submitted 2010-08-30; First posted 2010-09-02 (Estimated); Last update posted 2010-09-02 (Estimated); Status verified 2010-07

CONDITIONS: Humidity; Temperature
Keywords: Humidity; Temperature; Low Flow Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- humidity (Experimental)
  Interventions: Device: Datex Ohmeda excel anesthesia machine; Device: Datex Ohmeda Avance anesthesia work-station; Device: Drager Cato anesthesia work-station; Device: Drager Primus anesthesia work-station

INTERVENTIONS:
Device: Datex Ohmeda excel anesthesia machine — maintain one of following fresh gas flow, 1 or 4 L/min (nitrous oxide:oxygen =1:1) during 2 hour with using Datex Ohmeda excel anesthesia machine after draping complete
  Other Names: Excel
Device: Datex Ohmeda Avance anesthesia work-station — maintain one of following fresh gas flow, 0.5 or 1 or 4 L/min (nitrous oxide:oxygen =1:1) during 2 hour with using Datex Ohmeda Avance anesthesia machine after draping complete
  Other Names: Avance
Device: Drager Cato anesthesia work-station — maintain one of following fresh gas flow, 0.5 or 1 or 4 L/min (nitrous oxide:oxygen =1:1) during 2 hour with using Drager Cato anesthesia work-station after draping complete
  Other Names: Cato
Device: Drager Primus anesthesia work-station — maintain one of following fresh gas flow, 0.5 or 1 or 4 L/min (nitrous oxide:oxygen =1:1) during 2 hour with using Drager Primus anesthesia work-station after draping complete
  Other Names: Primus

SUMMARY:
The effects of preserving humidity and temperature by low flow anesthesia are different in each other anesthesia workstation.

DETAILED DESCRIPTION:
The fresh gas flow(FGF) is dry and cold in old fashioned anesthesia machine, especially at high folw (above 1 L/min). To the contrary, it has been assumed that the heat and humidity of FGF may be preserved using low FGF (below 1 L/min) during anesthesia or new anesthesia work station. However, it has not been proved yet. We hypothesized that the heat and moisture of FGF may be different in various FGF rate during anesthesia. In addition, it may be different in accordance to anesthesia work station. Therefore, we planed prospective observational study that will demonstrate that the difference of heat and moisture of FGF in different anesthesia work station (Excel; 1st generation anesthesia machine of Datex-Ohmeda Corp., Avance; 2nd generation anesthesia work station of Datex-Ohmeda Corp., Cato; 2nd generation generation anesthesia work station of Drager, Primus; 3rd generation generation anesthesia work station of Drager) and different FGF (0.5, 1, 4 L/min)

ELIGIBILITY:
Inclusion Criteria:

* patients who planned more than 2 hour operation under general anesthesia
* ASA class 1,2
* blood loss less than 500ml

Exclusion Criteria:

* acute/chronic cardiac or respiratory disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-09 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
absolute humidity at both limb of breathing circuit just distal portion of Y-piece | time point 1-11
  time point 1; base line value (fresh gas flow(FGF); 8L/min) time point 2; 5 mintues(min) after FGF change to predetermined level time point 3; 10 min after FGF change to predetermined level time point 4; 15 min after FGF change to predetermined level time point 5; 30 min after FGF change to predetermined level time point 6; 45 min after FGF change to predetermined level time point 7; 60 min time point 8; 75 min time point 9; 90 min time point 10; 105 min time point 11; 120 min

SECONDARY OUTCOMES:
patient body temperature(BT) | time point 1 -11
  measure BT using esophageal temperature probe each time points are same as primary outcome
temperature at both limb of breathing circuit just distal portion of Y-piece | time point 1- 11
  the time points are same as primary outcome

CONTACTS AND LOCATIONS:
Overall Officials: Seung Zhoo Yoon, Assist. P., Principal Investigator — Korea University Anam Hospital
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea